CLINICAL TRIAL: NCT00808067
Title: RELY-ABLE Long Term Multi-center Extension of Dabigatran Treatment in Patients With Atrial Fibrillation Who Completed the RE-LY Trial and a Cluster Randomised Trial to Assess the Effect of a Knowledge Translation Intervention on Patient Outcomes
Brief Title: RELY-ABLE Long Term Multi-center Extension of Dabigatran Treatment in Patients With Atrial Fibrillation Who Completed RE-LY Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1160.71; 2008-005248-17 (EudraCT Number: EudraCT)
Record Dates: First submitted 2008-12-12; First posted 2008-12-15 (Estimated); Results first posted 2014-04-08 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

ARMS (2):
- dabigatran dose 1 (Experimental): dabigatran high dose twice daily
  Interventions: Drug: dabigatran dose 1
- dabigatran dose 2 (Experimental): dabigatran low dose twice daily
  Interventions: Drug: dabigatran dose 2

INTERVENTIONS:
Drug: dabigatran dose 1 — dabigatran high dose twice daily
  Arms: dabigatran dose 1
Drug: dabigatran dose 2 — dabigatran low dose twice daily
  Arms: dabigatran dose 2

SUMMARY:
The purposes of this study are:

1. To evaluate the long-term safety of dabigatran etexilate
2. To assess the effect of a knowledge translation intervention on patient outcomes

ELIGIBILITY:
Inclusion criteria:

Participation in RE-LY, requires long term anticoagulation, provides written informed consent

Exclusion criteria:

Permanent discontinuation of dabigatran during RE-LY

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5897 (Actual)
Dates: Start 2008-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (567):
- United States (216):
  - 1160.71.0046 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 1160.71.0057 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 1160.71.0211 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 1160.71.0115 Boehringer Ingelheim Investigational Site, Mobile, Alabama
  - 1160.71.0104 Boehringer Ingelheim Investigational Site, Lake Havasu City, Arizona
  - 1160.71.0185 Boehringer Ingelheim Investigational Site, Tucson, Arizona
  - 1160.71.0038 Boehringer Ingelheim Investigational Site, Hot Springs, Arkansas
  - 1160.71.0302 Boehringer Ingelheim Investigational Site, Jonesboro, Arkansas
  - 1160.71.0191 Boehringer Ingelheim Investigational Site, Little Rock, Arkansas
  - 1160.71.0213 Boehringer Ingelheim Investigational Site, Little Rock, Arkansas
  - 1160.71.0441 Boehringer Ingelheim Investigational Site, Carmichael, California
  - 1160.71.0333 Boehringer Ingelheim Investigational Site, Fullerton, California
  - 1160.71.0384 Boehringer Ingelheim Investigational Site, La Jolla, California
  - 1160.71.0246 Boehringer Ingelheim Investigational Site, Lancaster, California
  - 1160.71.0070 Boehringer Ingelheim Investigational Site, Merced, California
  - 1160.71.0349 Boehringer Ingelheim Investigational Site, Oakland, California
  - 1160.71.0016 Boehringer Ingelheim Investigational Site, Oceanside, California
  - 1160.71.0459 Boehringer Ingelheim Investigational Site, Pasadena, California
  - 1160.71.0270 Boehringer Ingelheim Investigational Site, Poway, California
  - 1160.71.0135 Boehringer Ingelheim Investigational Site, Riverside, California
  - 1160.71.0300 Boehringer Ingelheim Investigational Site, Sacramento, California
  - 1160.71.0284 Boehringer Ingelheim Investigational Site, San Diego, California
  - 1160.71.0379 Boehringer Ingelheim Investigational Site, Walnut Creek, California
  - 1160.71.0321 Boehringer Ingelheim Investigational Site, Colorado Springs, Colorado
  - 1160.71.0449 Boehringer Ingelheim Investigational Site, Colorado Springs, Colorado
  - 1160.71.0360 Boehringer Ingelheim Investigational Site, Denver, Colorado
  - 1160.71.0413 Boehringer Ingelheim Investigational Site, Denver, Colorado
  - 1160.71.0362 Boehringer Ingelheim Investigational Site, Fort Collins, Colorado
  - 1160.71.0278 Boehringer Ingelheim Investigational Site, Bridgeport, Connecticut
  - 1160.71.0482 Boehringer Ingelheim Investigational Site, Guilford, Connecticut
  - 1160.71.0382 Boehringer Ingelheim Investigational Site, Boynton Beach, Florida
  - 1160.71.0056 Boehringer Ingelheim Investigational Site, Brandon, Florida
  - 1160.71.0296 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 1160.71.0327 Boehringer Ingelheim Investigational Site, Coral Springs, Florida
  - 1160.71.0376 Boehringer Ingelheim Investigational Site, Daytona Beach, Florida
  - 1160.71.0074 Boehringer Ingelheim Investigational Site, Fort Myers, Florida
  - 1160.71.0089 Boehringer Ingelheim Investigational Site, Jacksonville, Florida
  - 1160.71.0232 Boehringer Ingelheim Investigational Site, Jacksonville, Florida
  - 1160.71.0427 Boehringer Ingelheim Investigational Site, Jacksonville, Florida
  - 1160.71.0012 Boehringer Ingelheim Investigational Site, Lakeland, Florida
  - 1160.71.0034 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1160.71.0227 Boehringer Ingelheim Investigational Site, Orlando, Florida
  - 1160.71.0095 Boehringer Ingelheim Investigational Site, Ormond Beach, Florida
  - 1160.71.0037 Boehringer Ingelheim Investigational Site, Pensacola, Florida
  - 1160.71.0137 Boehringer Ingelheim Investigational Site, Port Charlotte, Florida
  - 1160.71.0417 Boehringer Ingelheim Investigational Site, Port Charlotte, Florida
  - 1160.71.0332 Boehringer Ingelheim Investigational Site, Rockledge, Florida
  - 1160.71.0385 Boehringer Ingelheim Investigational Site, Sarasota, Florida
  - 1160.71.0015 Boehringer Ingelheim Investigational Site, St. Petersburg, Florida
  - 1160.71.0339 Boehringer Ingelheim Investigational Site, St. Petersburg, Florida
  - 1160.71.0019 Boehringer Ingelheim Investigational Site, Vero Beach, Florida
  - 1160.71.0159 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 1160.71.0021 Boehringer Ingelheim Investigational Site, Augusta, Georgia
  - 1160.71.0161 Boehringer Ingelheim Investigational Site, Conyers, Georgia
  - 1160.71.0218 Boehringer Ingelheim Investigational Site, Cicero, Illinois
  - 1160.71.0438 Boehringer Ingelheim Investigational Site, Maywood, Illinois
  - 1160.71.0331 Boehringer Ingelheim Investigational Site, Melrose Park, Illinois
  - 1160.71.0364 Boehringer Ingelheim Investigational Site, Normal, Illinois
  - 1160.71.0109 Boehringer Ingelheim Investigational Site, North Chicago, Illinois
  - 1160.71.0152 Boehringer Ingelheim Investigational Site, Oak Lawn, Illinois
  - 1160.71.0198 Boehringer Ingelheim Investigational Site, Rockford, Illinois
  - 1160.71.0433 Boehringer Ingelheim Investigational Site, Winfield, Illinois
  - 1160.71.0377 Boehringer Ingelheim Investigational Site, Fort Wayne, Indiana
  - 1160.71.0288 Boehringer Ingelheim Investigational Site, Indianapolis, Indiana
  - 1160.71.0352 Boehringer Ingelheim Investigational Site, Indianapolis, Indiana
  - 1160.71.0436 Boehringer Ingelheim Investigational Site, Indianapolis, Indiana
  - 1160.71.0235 Boehringer Ingelheim Investigational Site, South Bend, Indiana
  - 1160.71.0268 Boehringer Ingelheim Investigational Site, Dubuque, Iowa
  - 1160.71.0001 Boehringer Ingelheim Investigational Site, West Des Moines, Iowa
  - 1160.71.0357 Boehringer Ingelheim Investigational Site, West Des Moines, Iowa
  - 1160.71.0422 Boehringer Ingelheim Investigational Site, Lexington, Kentucky
  - 1160.71.0178 Boehringer Ingelheim Investigational Site, Louisville, Kentucky
  - 1160.71.0397 Boehringer Ingelheim Investigational Site, Louisville, Kentucky
  - 1160.71.0310 Boehringer Ingelheim Investigational Site, Owensboro, Kentucky
  - 1160.71.0144 Boehringer Ingelheim Investigational Site, Baton Rouge, Louisiana
  - 1160.71.0018 Boehringer Ingelheim Investigational Site, Lafayette, Louisiana
  - 1160.71.0132 Boehringer Ingelheim Investigational Site, New Iberia, Louisiana
  - 1160.71.0096 Boehringer Ingelheim Investigational Site, Auburn, Maine
  - 1160.71.0114 Boehringer Ingelheim Investigational Site, Annapolis, Maryland
  - 1160.71.0023 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 1160.71.0047 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 1160.71.0079 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 1160.71.0186 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 1160.71.0194 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 1160.71.0255 Boehringer Ingelheim Investigational Site, Bel Air, Maryland
  - 1160.71.0398 Boehringer Ingelheim Investigational Site, Columbia, Maryland
  - 1160.71.0177 Boehringer Ingelheim Investigational Site, Rockville, Maryland
  - 1160.71.0073 Boehringer Ingelheim Investigational Site, Salisbury, Maryland
  - 1160.71.0207 Boehringer Ingelheim Investigational Site, Salisbury, Maryland
  - 1160.71.0196 Boehringer Ingelheim Investigational Site, Takoma Park, Maryland
  - 1160.71.0187 Boehringer Ingelheim Investigational Site, Towson, Maryland
  - 1160.71.0052 Boehringer Ingelheim Investigational Site, Westminster, Maryland
  - 1160.71.0443 Boehringer Ingelheim Investigational Site, Haverhill, Massachusetts
  - 1160.71.0452 Boehringer Ingelheim Investigational Site, Haverhill, Massachusetts
  - 1160.71.0029 Boehringer Ingelheim Investigational Site, Natick, Massachusetts
  - 1160.71.0003 Boehringer Ingelheim Investigational Site, North Dartmouth, Massachusetts
  - 1160.71.0308 Boehringer Ingelheim Investigational Site, Worcester, Massachusetts
  - 1160.71.0154 Boehringer Ingelheim Investigational Site, Grand Blanc, Michigan
  - 1160.71.0205 Boehringer Ingelheim Investigational Site, Lapeer, Michigan
  - 1160.71.0279 Boehringer Ingelheim Investigational Site, Muskegon, Michigan
  - 1160.71.0445 Boehringer Ingelheim Investigational Site, Petoskey, Michigan
  - 1160.71.0274 Boehringer Ingelheim Investigational Site, Rochester Hills, Michigan
  - 1160.71.0165 Boehringer Ingelheim Investigational Site, Saginaw, Michigan
  - 1160.71.0020 Boehringer Ingelheim Investigational Site, Troy, Michigan
  - 1160.71.0188 Boehringer Ingelheim Investigational Site, Ypsilanti, Michigan
  - 1160.71.0202 Boehringer Ingelheim Investigational Site, Minneapolis, Minnesota
  - 1160.71.0101 Boehringer Ingelheim Investigational Site, Saint Paul, Minnesota
  - 1160.71.0086 Boehringer Ingelheim Investigational Site, Gulfport, Mississippi
  - 1160.71.0119 Boehringer Ingelheim Investigational Site, Tupelo, Mississippi
  - 1160.71.0055 Boehringer Ingelheim Investigational Site, Columbia, Missouri
  - 1160.71.0257 Boehringer Ingelheim Investigational Site, Kansas City, Missouri
  - 1160.71.0336 Boehringer Ingelheim Investigational Site, Saint Charles, Missouri
  - 1160.71.0249 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 1160.71.0027 Boehringer Ingelheim Investigational Site, Kalispell, Montana
  - 1160.71.0110 Boehringer Ingelheim Investigational Site, Omaha, Nebraska
  - 1160.71.0346 Boehringer Ingelheim Investigational Site, Henderson, Nevada
  - 1160.71.0430 Boehringer Ingelheim Investigational Site, Las Vegas, Nevada
  - 1160.71.0142 Boehringer Ingelheim Investigational Site, Browns Mills, New Jersey
  - 1160.71.0221 Boehringer Ingelheim Investigational Site, Cherry Hill, New Jersey
  - 1160.71.0248 Boehringer Ingelheim Investigational Site, Flemington, New Jersey
  - 1160.71.0478 Boehringer Ingelheim Investigational Site, Oakland, New Jersey
  - 1160.71.0392 Boehringer Ingelheim Investigational Site, Ocean City, New Jersey
  - 1160.71.0254 Boehringer Ingelheim Investigational Site, Westwood, New Jersey
  - 1160.71.0472 Boehringer Ingelheim Investigational Site, Woodland Park, New Jersey
  - 1160.71.0476 Boehringer Ingelheim Investigational Site, Albany, New York
  - 1160.71.0044 Boehringer Ingelheim Investigational Site, Cortlandt Manor, New York
  - 1160.71.0229 Boehringer Ingelheim Investigational Site, Mineola, New York
  - 1160.71.0451 Boehringer Ingelheim Investigational Site, Mineola, New York
  - 1160.71.0183 Boehringer Ingelheim Investigational Site, New Rochelle, New York
  - 1160.71.0210 Boehringer Ingelheim Investigational Site, Northport, New York
  - 1160.71.0075 Boehringer Ingelheim Investigational Site, Poughkeepsie, New York
  - 1160.71.0113 Boehringer Ingelheim Investigational Site, The Bronx, New York
  - 1160.71.0281 Boehringer Ingelheim Investigational Site, The Bronx, New York
  - 1160.71.0414 Boehringer Ingelheim Investigational Site, Troy, New York
  - 1160.71.0356 Boehringer Ingelheim Investigational Site, Watertown, New York
  - 1160.71.0064 Boehringer Ingelheim Investigational Site, Yonkers, New York
  - 1160.71.0353 Boehringer Ingelheim Investigational Site, Asheville, North Carolina
  - 1160.71.0080 Boehringer Ingelheim Investigational Site, Charlotte, North Carolina
  - 1160.71.0350 Boehringer Ingelheim Investigational Site, Gastonia, North Carolina
  - 1160.71.0173 Boehringer Ingelheim Investigational Site, High Point, North Carolina
  - 1160.71.0006 Boehringer Ingelheim Investigational Site, Pinehurst, North Carolina
  - 1160.71.0002 Boehringer Ingelheim Investigational Site, Statesville, North Carolina
  - 1160.71.0069 Boehringer Ingelheim Investigational Site, Statesville, North Carolina
  - 1160.71.0102 Boehringer Ingelheim Investigational Site, Grand Forks, North Dakota
  - 1160.71.0222 Boehringer Ingelheim Investigational Site, Jamestown, North Dakota
  - 1160.71.0203 Boehringer Ingelheim Investigational Site, Akron, Ohio
  - 1160.71.0434 Boehringer Ingelheim Investigational Site, Canal Fulton, Ohio
  - 1160.71.0402 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1160.71.0426 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1160.71.0479 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1160.71.0263 Boehringer Ingelheim Investigational Site, Cleveland, Ohio
  - 1160.71.0480 Boehringer Ingelheim Investigational Site, Cleveland, Ohio
  - 1160.71.0267 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 1160.71.0035 Boehringer Ingelheim Investigational Site, Dayton, Ohio
  - 1160.71.0150 Boehringer Ingelheim Investigational Site, Fairview Park, Ohio
  - 1160.71.0201 Boehringer Ingelheim Investigational Site, Kettering, Ohio
  - 1160.71.0223 Boehringer Ingelheim Investigational Site, Lorain, Ohio
  - 1160.71.0214 Boehringer Ingelheim Investigational Site, Lyndhurst, Ohio
  - 1160.71.0275 Boehringer Ingelheim Investigational Site, Sandusky, Ohio
  - 1160.71.0103 Boehringer Ingelheim Investigational Site, Westlake, Ohio
  - 1160.71.0435 Boehringer Ingelheim Investigational Site, Tulsa, Oklahoma
  - 1160.71.0139 Boehringer Ingelheim Investigational Site, Corvallis, Oregon
  - 1160.71.0325 Boehringer Ingelheim Investigational Site, Eugene, Oregon
  - 1160.71.0133 Boehringer Ingelheim Investigational Site, Springfield, Oregon
  - 1160.71.0301 Boehringer Ingelheim Investigational Site, Allentown, Pennsylvania
  - 1160.71.0295 Boehringer Ingelheim Investigational Site, Camp Hill, Pennsylvania
  - 1160.71.0294 Boehringer Ingelheim Investigational Site, Hershey, Pennsylvania
  - 1160.71.0369 Boehringer Ingelheim Investigational Site, Jenkintown, Pennsylvania
  - 1160.71.0431 Boehringer Ingelheim Investigational Site, Lancaster, Pennsylvania
  - 1160.71.0168 Boehringer Ingelheim Investigational Site, Langhorne, Pennsylvania
  - 1160.71.0293 Boehringer Ingelheim Investigational Site, Meadowbrook, Pennsylvania
  - 1160.71.0394 Boehringer Ingelheim Investigational Site, Norristown, Pennsylvania
  - 1160.71.0466 Boehringer Ingelheim Investigational Site, Pittsburgh, Pennsylvania
  - 1160.71.0208 Boehringer Ingelheim Investigational Site, Sellersville, Pennsylvania
  - 1160.71.0465 Boehringer Ingelheim Investigational Site, Uniontown, Pennsylvania
  - 1160.71.0032 Boehringer Ingelheim Investigational Site, Wynnewood, Pennsylvania
  - 1160.71.0067 Boehringer Ingelheim Investigational Site, Wyomissing, Pennsylvania
  - 1160.71.0007 Boehringer Ingelheim Investigational Site, Beaufort, South Carolina
  - 1160.71.0383 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 1160.71.0313 Boehringer Ingelheim Investigational Site, Greenville, South Carolina
  - 1160.71.0166 Boehringer Ingelheim Investigational Site, Spartanburg, South Carolina
  - 1160.71.0008 Boehringer Ingelheim Investigational Site, Summerville, South Carolina
  - 1160.71.0084 Boehringer Ingelheim Investigational Site, Chattanooga, Tennessee
  - 1160.71.0474 Boehringer Ingelheim Investigational Site, Clinton, Tennessee
  - 1160.71.0062 Boehringer Ingelheim Investigational Site, Germantown, Tennessee
  - 1160.71.0370 Boehringer Ingelheim Investigational Site, Johnson City, Tennessee
  - 1160.71.0395 Boehringer Ingelheim Investigational Site, Nashville, Tennessee
  - 1160.71.0129 Boehringer Ingelheim Investigational Site, Austin, Texas
  - 1160.71.0410 Boehringer Ingelheim Investigational Site, Austin, Texas
  - 1160.71.0156 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1160.71.0315 Boehringer Ingelheim Investigational Site, Fort Worth, Texas
  - 1160.71.0447 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1160.71.0483 Boehringer Ingelheim Investigational Site, Killeen, Texas
  - 1160.71.0335 Boehringer Ingelheim Investigational Site, Lubbock, Texas
  - 1160.71.0269 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1160.71.0307 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1160.71.0285 Boehringer Ingelheim Investigational Site, San Marcos, Texas
  - 1160.71.0367 Boehringer Ingelheim Investigational Site, Tyler, Texas
  - 1160.71.0453 Boehringer Ingelheim Investigational Site, Charlottesville, Virginia
  - 1160.71.0053 Boehringer Ingelheim Investigational Site, Chesapeake, Virginia
  - 1160.71.0428 Boehringer Ingelheim Investigational Site, Fredericksburg, Virginia
  - 1160.71.0311 Boehringer Ingelheim Investigational Site, Harrisonburg, Virginia
  - 1160.71.0292 Boehringer Ingelheim Investigational Site, Newport News, Virginia
  - 1160.71.0220 Boehringer Ingelheim Investigational Site, Salem, Virginia
  - 1160.71.0224 Boehringer Ingelheim Investigational Site, Suffolk, Virginia
  - 1160.71.0317 Boehringer Ingelheim Investigational Site, Winchester, Virginia
  - 1160.71.0050 Boehringer Ingelheim Investigational Site, Bellingham, Washington
  - 1160.71.0040 Boehringer Ingelheim Investigational Site, Burien, Washington
  - 1160.71.0250 Boehringer Ingelheim Investigational Site, Spokane, Washington
  - 1160.71.0256 Boehringer Ingelheim Investigational Site, Tacoma, Washington
  - 1160.71.0024 Boehringer Ingelheim Investigational Site, Wenatchee, Washington
  - 1160.71.0169 Boehringer Ingelheim Investigational Site, Clarksburg, West Virginia
  - 1160.71.0365 Boehringer Ingelheim Investigational Site, Huntington, West Virginia
  - 1160.71.0099 Boehringer Ingelheim Investigational Site, Madison, Wisconsin
  - 1160.71.0072 Boehringer Ingelheim Investigational Site, Milwaukee, Wisconsin
  - 1160.71.0461 Boehringer Ingelheim Investigational Site, Milwaukee, Wisconsin
- Australia (7):
  - 1160.71.0508 Boehringer Ingelheim Investigational Site, Coffs Harbour, New South Wales
  - 1160.71.0510 Boehringer Ingelheim Investigational Site, Gosford, New South Wales
  - 1160.71.0506 Boehringer Ingelheim Investigational Site, Milton, Queensland
  - 1160.71.0509 Boehringer Ingelheim Investigational Site, Ashford, South Australia
  - 1160.71.0507 Boehringer Ingelheim Investigational Site, Launceston, Tasmania
  - 1160.71.0504 Boehringer Ingelheim Investigational Site, Box Hill, Victoria
  - 1160.71.0501 Boehringer Ingelheim Investigational Site, Geelong, Victoria
- Austria (8):
  - 1160.71.0543 Boehringer Ingelheim Investigational Site, Graz
  - 1160.71.0549 Boehringer Ingelheim Investigational Site, Linz
  - 1160.71.0541 Boehringer Ingelheim Investigational Site, Vienna
  - 1160.71.0542 Boehringer Ingelheim Investigational Site, Vienna
  - 1160.71.0545 Boehringer Ingelheim Investigational Site, Vienna
  - 1160.71.0547 Boehringer Ingelheim Investigational Site, Vienna
  - 1160.71.0548 Boehringer Ingelheim Investigational Site, Vienna
  - 1160.71.0550 Boehringer Ingelheim Investigational Site, Wiener Neustadt
- Belgium (17):
  - 1160.71.0564 Boehringer Ingelheim Investigational Site, Aalst
  - 1160.71.0572 Boehringer Ingelheim Investigational Site, Brasschaat
  - 1160.71.0571 Boehringer Ingelheim Investigational Site, Brussels
  - 1160.71.0581 Boehringer Ingelheim Investigational Site, Brussels
  - 1160.71.0585 Boehringer Ingelheim Investigational Site, Brussels
  - 1160.71.0563 Boehringer Ingelheim Investigational Site, Edegem
  - 1160.71.0578 Boehringer Ingelheim Investigational Site, Genk
  - 1160.71.0587 Boehringer Ingelheim Investigational Site, Genk
  - 1160.71.0574 Boehringer Ingelheim Investigational Site, Ghent
  - 1160.71.0588 Boehringer Ingelheim Investigational Site, Gilly
  - 1160.71.0568 Boehringer Ingelheim Investigational Site, Hasselt
  - 1160.71.0561 Boehringer Ingelheim Investigational Site, Leuven
  - 1160.71.0579 Boehringer Ingelheim Investigational Site, Liège
  - 1160.71.0567 Boehringer Ingelheim Investigational Site, Ostend
  - 1160.71.0570 Boehringer Ingelheim Investigational Site, Roeselare
  - 1160.71.0566 Boehringer Ingelheim Investigational Site, Tienen
  - 1160.71.0562 Boehringer Ingelheim Investigational Site, Turnhout
- Brazil (7):
  - 1160.71.0644 Boehringer Ingelheim Investigational Site, Campinas
  - 1160.71.0650 Boehringer Ingelheim Investigational Site, Curitiba
  - 1160.71.0651 Boehringer Ingelheim Investigational Site, Curitiba
  - 1160.71.0652 Boehringer Ingelheim Investigational Site, Goiânia
  - 1160.71.0646 Boehringer Ingelheim Investigational Site, Sao Jose Do Riio Preto
  - 1160.71.0647 Boehringer Ingelheim Investigational Site, São José do Rio Preto
  - 1160.71.0643 Boehringer Ingelheim Investigational Site, São Paulo
- Bulgaria (7):
  - 1160.71.0620 Boehringer Ingelheim Investigational Site, Pleven
  - 1160.71.0611 Boehringer Ingelheim Investigational Site, Sofia
  - 1160.71.0612 Boehringer Ingelheim Investigational Site, Sofia
  - 1160.71.0615 Boehringer Ingelheim Investigational Site, Sofia
  - 1160.71.0617 Boehringer Ingelheim Investigational Site, Sofia
  - 1160.71.0618 Boehringer Ingelheim Investigational Site, Sofia
  - 1160.71.0625 Boehringer Ingelheim Investigational Site, Sofia
- Canada (40):
  - 1160.71.0694 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 1160.71.0696 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 1160.71.0680 Boehringer Ingelheim Investigational Site, Coquitlam, British Columbia
  - 1160.71.0712 Boehringer Ingelheim Investigational Site, Coquitlam, British Columbia
  - 1160.71.0706 Boehringer Ingelheim Investigational Site, Kelowna, British Columbia
  - 1160.71.0725 Boehringer Ingelheim Investigational Site, Nanaimo, British Columbia
  - 1160.71.0691 Boehringer Ingelheim Investigational Site, New Westminster, British Columbia
  - 1160.71.0714 Boehringer Ingelheim Investigational Site, Victoria, British Columbia
  - 1160.71.0701 Boehringer Ingelheim Investigational Site, Portage la Prairie, Manitoba
  - 1160.71.0703 Boehringer Ingelheim Investigational Site, Halifax, Nova Scotia
  - 1160.71.0674 Boehringer Ingelheim Investigational Site, Burlington, Ontario
  - 1160.71.0702 Boehringer Ingelheim Investigational Site, Cambridge, Ontario
  - 1160.71.0720 Boehringer Ingelheim Investigational Site, Cambridge, Ontario
  - 1160.71.0715 Boehringer Ingelheim Investigational Site, Greater Sudbury, Ontario
  - 1160.71.0692 Boehringer Ingelheim Investigational Site, Grimsby, Ontario
  - 1160.71.0697 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1160.71.0710 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1160.71.0719 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1160.71.0721 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1160.71.0708 Boehringer Ingelheim Investigational Site, Mississauga, Ontario
  - 1160.71.0688 Boehringer Ingelheim Investigational Site, Newmarket, Ontario
  - 1160.71.0672 Boehringer Ingelheim Investigational Site, Oshawa, Ontario
  - 1160.71.0687 Boehringer Ingelheim Investigational Site, Ottawa, Ontario
  - 1160.71.0679 Boehringer Ingelheim Investigational Site, Scarborough Village, Ontario
  - 1160.71.0723 Boehringer Ingelheim Investigational Site, Scarborough Village, Ontario
  - 1160.71.0690 Boehringer Ingelheim Investigational Site, Thunder Bay, Ontario
  - 1160.71.0684 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1160.71.0718 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1160.71.0686 Boehringer Ingelheim Investigational Site, Windsor, Ontario
  - 1160.71.0683 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1160.71.0705 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1160.71.0709 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1160.71.0716 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1160.71.0700 Boehringer Ingelheim Investigational Site, Québec, Quebec
  - 1160.71.0717 Boehringer Ingelheim Investigational Site, Québec, Quebec
  - 1160.71.0713 Boehringer Ingelheim Investigational Site, Saint George-de-Beauce, Quebec
  - 1160.71.0699 Boehringer Ingelheim Investigational Site, Saint-Charles-Borromée, Quebec
  - 1160.71.0675 Boehringer Ingelheim Investigational Site, Saint-Hyacinthe, Quebec
  - 1160.71.0673 Boehringer Ingelheim Investigational Site, Saskatoon, Saskatchewan
  - 1160.71.0678 Boehringer Ingelheim Investigational Site, Saskatoon, Saskatchewan
- China (11):
  - 1160.71.0771 Boehringer Ingelheim Investigational Site, Beijing
  - 1160.71.0772 Boehringer Ingelheim Investigational Site, Beijing
  - 1160.71.0773 Boehringer Ingelheim Investigational Site, Beijing
  - 1160.71.0774 Boehringer Ingelheim Investigational Site, Beijing
  - 1160.71.0776 Boehringer Ingelheim Investigational Site, Haerbin
  - 1160.71.0784 Boehringer Ingelheim Investigational Site, Hangzhou
  - 1160.71.0778 Boehringer Ingelheim Investigational Site, Qingdao
  - 1160.71.0781 Boehringer Ingelheim Investigational Site, Shanghai
  - 1160.71.0782 Boehringer Ingelheim Investigational Site, Shanghai
  - 1160.71.0777 Boehringer Ingelheim Investigational Site, Shenyang
  - 1160.71.0780 Boehringer Ingelheim Investigational Site, Shijiazhuang
- Czechia (9):
  - 1160.71.0816 Boehringer Ingelheim Investigational Site, Modřice
  - 1160.71.0820 Boehringer Ingelheim Investigational Site, Ostrava
  - 1160.71.0818 Boehringer Ingelheim Investigational Site, Pardubice
  - 1160.71.0814 Boehringer Ingelheim Investigational Site, Plzen-Bory
  - 1160.71.0811 Boehringer Ingelheim Investigational Site, Prague
  - 1160.71.0812 Boehringer Ingelheim Investigational Site, Prague
  - 1160.71.0813 Boehringer Ingelheim Investigational Site, Prague
  - 1160.71.0817 Boehringer Ingelheim Investigational Site, Příbram
  - 1160.71.0819 Boehringer Ingelheim Investigational Site, Ústí nad Orlicí
- Denmark (11):
  - 1160.71.0837 Boehringer Ingelheim Investigational Site, Aalborg
  - 1160.71.0835 Boehringer Ingelheim Investigational Site, Aarhus C
  - 1160.71.0833 Boehringer Ingelheim Investigational Site, Elsinore
  - 1160.71.0838 Boehringer Ingelheim Investigational Site, Frederikssund
  - 1160.71.0834 Boehringer Ingelheim Investigational Site, Herlev
  - 1160.71.0841 Boehringer Ingelheim Investigational Site, Horsens
  - 1160.71.0832 Boehringer Ingelheim Investigational Site, Hvidovre
  - 1160.71.0840 Boehringer Ingelheim Investigational Site, Køge
  - 1160.71.0831 Boehringer Ingelheim Investigational Site, Odense
  - 1160.71.0839 Boehringer Ingelheim Investigational Site, Roskilde
  - 1160.71.0836 Boehringer Ingelheim Investigational Site, Svendborg
- Finland (6):
  - 1160.71.0851 Boehringer Ingelheim Investigational Site, Helsinki
  - 1160.71.0859 Boehringer Ingelheim Investigational Site, Jyväskylä
  - 1160.71.0854 Boehringer Ingelheim Investigational Site, Oulu
  - 1160.71.0858 Boehringer Ingelheim Investigational Site, Pori
  - 1160.71.0852 Boehringer Ingelheim Investigational Site, Tampere
  - 1160.71.0853 Boehringer Ingelheim Investigational Site, Turku
- France (26):
  - 1160.71.875A Boehringer Ingelheim Investigational Site, Abbeville
  - 1160.71.882D Boehringer Ingelheim Investigational Site, Angers
  - 1160.71.882G Boehringer Ingelheim Investigational Site, Angers
  - 1160.71.879F Boehringer Ingelheim Investigational Site, Besle Sur Vilaine
  - 1160.71.882K Boehringer Ingelheim Investigational Site, Château-Gontier
  - 1160.71.887A Boehringer Ingelheim Investigational Site, Cholet
  - 1160.71.879C Boehringer Ingelheim Investigational Site, Derval
  - 1160.71.882H Boehringer Ingelheim Investigational Site, Feneu
  - 1160.71.888A Boehringer Ingelheim Investigational Site, Grenoble Cédex 9
  - 1160.71.879B Boehringer Ingelheim Investigational Site, La Chapelle-sur-Erdre
  - 1160.71.874A Boehringer Ingelheim Investigational Site, Langres
  - 1160.71.884A Boehringer Ingelheim Investigational Site, Laval
  - 1160.71.880B Boehringer Ingelheim Investigational Site, Le Mesnil En Valée
  - 1160.71.880A Boehringer Ingelheim Investigational Site, Mûrs-Erigné
  - 1160.71.879A Boehringer Ingelheim Investigational Site, Nantes
  - 1160.71.879H Boehringer Ingelheim Investigational Site, Nantes
  - 1160.71.879S Boehringer Ingelheim Investigational Site, Nantes
  - 1160.71.880J Boehringer Ingelheim Investigational Site, Parçay-les-Pins
  - 1160.71.871A Boehringer Ingelheim Investigational Site, Paris
  - 1160.71.879E Boehringer Ingelheim Investigational Site, Saint-Aubin-des-Châteaux
  - 1160.71.880D Boehringer Ingelheim Investigational Site, Segré
  - 1160.71.882A Boehringer Ingelheim Investigational Site, Tiercé
  - 1160.71.882B Boehringer Ingelheim Investigational Site, Tiercé
  - 1160.71.882C Boehringer Ingelheim Investigational Site, Tiercé
  - 1160.71.879G Boehringer Ingelheim Investigational Site, Vieillevigne
  - 1160.71.880E Boehringer Ingelheim Investigational Site, Vihiers
- Germany (17):
  - 1160.71.0932 Boehringer Ingelheim Investigational Site, Berlin
  - 1160.71.0948 Boehringer Ingelheim Investigational Site, Berlin
  - 1160.71.0962 Boehringer Ingelheim Investigational Site, Berlin
  - 1160.71.0940 Boehringer Ingelheim Investigational Site, Bochum
  - 1160.71.0963 Boehringer Ingelheim Investigational Site, Cologne
  - 1160.71.0972 Boehringer Ingelheim Investigational Site, Dortmund
  - 1160.71.0934 Boehringer Ingelheim Investigational Site, Essen
  - 1160.71.0931 Boehringer Ingelheim Investigational Site, Frankfurt am Main
  - 1160.71.0943 Boehringer Ingelheim Investigational Site, Heidelberg
  - 1160.71.0946 Boehringer Ingelheim Investigational Site, Lahr
  - 1160.71.0944 Boehringer Ingelheim Investigational Site, Limburg
  - 1160.71.0951 Boehringer Ingelheim Investigational Site, Mainz
  - 1160.71.0933 Boehringer Ingelheim Investigational Site, Mannheim
  - 1160.71.0945 Boehringer Ingelheim Investigational Site, Mannheim
  - 1160.71.0970 Boehringer Ingelheim Investigational Site, Mannheim
  - 1160.71.0937 Boehringer Ingelheim Investigational Site, Witten
  - 1160.71.0966 Boehringer Ingelheim Investigational Site, Wuppertal
- Greece (6):
  - 1160.71.0901 Boehringer Ingelheim Investigational Site, Athens
  - 1160.71.0914 Boehringer Ingelheim Investigational Site, Kalamaria-Thessaloniki
  - 1160.71.0904 Boehringer Ingelheim Investigational Site, Larissa
  - 1160.71.0910 Boehringer Ingelheim Investigational Site, Thebes
  - 1160.71.0903 Boehringer Ingelheim Investigational Site, Trikala
  - 1160.71.0905 Boehringer Ingelheim Investigational Site, Voula - Athens
- Hong Kong (2):
  - 1160.71.1003 Boehringer Ingelheim Investigational Site, Kowloon
  - 1160.71.1004 Boehringer Ingelheim Investigational Site, Kowloon
- Hungary (9):
  - 1160.71.1011 Boehringer Ingelheim Investigational Site, Budapest
  - 1160.71.1012 Boehringer Ingelheim Investigational Site, Budapest
  - 1160.71.1013 Boehringer Ingelheim Investigational Site, Budapest
  - 1160.71.1014 Boehringer Ingelheim Investigational Site, Budapest
  - 1160.71.1015 Boehringer Ingelheim Investigational Site, Budapest
  - 1160.71.1016 Boehringer Ingelheim Investigational Site, Budapest
  - 1160.71.1020 Boehringer Ingelheim Investigational Site, Gyöngyös
  - 1160.71.1017 Boehringer Ingelheim Investigational Site, Komárom
  - 1160.71.1018 Boehringer Ingelheim Investigational Site, Pécs
- India (13):
  - 1160.71.1057 Boehringer Ingelheim Investigational Site, Ahmedabad
  - 1160.71.1056 Boehringer Ingelheim Investigational Site, Ahmedabad-52
  - 1160.71.1065 Boehringer Ingelheim Investigational Site, Bangalore
  - 1160.71.1062 Boehringer Ingelheim Investigational Site, Hyderabad
  - 1160.71.1073 Boehringer Ingelheim Investigational Site, Jaipur, Rajasthan
  - 1160.71.1067 Boehringer Ingelheim Investigational Site, Kerala
  - 1160.71.1068 Boehringer Ingelheim Investigational Site, Kottayam
  - 1160.71.1055 Boehringer Ingelheim Investigational Site, Lucknow, Uttar Pradesh
  - 1160.71.1051 Boehringer Ingelheim Investigational Site, Ludhiana
  - 1160.71.1072 Boehringer Ingelheim Investigational Site, Mysore
  - 1160.71.1059 Boehringer Ingelheim Investigational Site, Nagpur-12
  - 1160.71.1052 Boehringer Ingelheim Investigational Site, New Delhi
  - 1160.71.1070 Boehringer Ingelheim Investigational Site, Pune, Maharashtra
- Israel (26):
  - 1160.71.1110 Boehringer Ingelheim Investigational Site, Afula
  - 1160.71.1121 Boehringer Ingelheim Investigational Site, Afula
  - 1160.71.1111 Boehringer Ingelheim Investigational Site, Ashkelon
  - 1160.71.1117 Boehringer Ingelheim Investigational Site, Giv‘atayim
  - 1160.71.1112 Boehringer Ingelheim Investigational Site, Hadera
  - 1160.71.1091 Boehringer Ingelheim Investigational Site, Haifa
  - 1160.71.1113 Boehringer Ingelheim Investigational Site, Haifa
  - 1160.71.1114 Boehringer Ingelheim Investigational Site, Haifa
  - 1160.71.1116 Boehringer Ingelheim Investigational Site, Haifa
  - 1160.71.1118 Boehringer Ingelheim Investigational Site, Haifa
  - 1160.71.1105 Boehringer Ingelheim Investigational Site, Holon
  - 1160.71.1101 Boehringer Ingelheim Investigational Site, Jerusalem
  - 1160.71.1104 Boehringer Ingelheim Investigational Site, Jerusalem
  - 1160.71.1106 Boehringer Ingelheim Investigational Site, Jerusalem
  - 1160.71.1119 Boehringer Ingelheim Investigational Site, Kfar Saba
  - 1160.71.1096 Boehringer Ingelheim Investigational Site, Petah Tikva
  - 1160.71.1093 Boehringer Ingelheim Investigational Site, Ramat Gan
  - 1160.71.1094 Boehringer Ingelheim Investigational Site, Ramat Gan
  - 1160.71.1095 Boehringer Ingelheim Investigational Site, Ramat Gan
  - 1160.71.1100 Boehringer Ingelheim Investigational Site, Rehovot
  - 1160.71.1103 Boehringer Ingelheim Investigational Site, Safed
  - 1160.71.1107 Boehringer Ingelheim Investigational Site, Tel Aviv
  - 1160.71.1108 Boehringer Ingelheim Investigational Site, Tel Aviv
  - 1160.71.1109 Boehringer Ingelheim Investigational Site, Tel Aviv
  - 1160.71.1120 Boehringer Ingelheim Investigational Site, Tel Aviv
  - 1160.71.1122 Boehringer Ingelheim Investigational Site, Tel Aviv
- Italy (3):
  - 1160.71.1169 Boehringer Ingelheim Investigational Site, Arezzo
  - 1160.71.1172 Boehringer Ingelheim Investigational Site, Ascoli Piceno
  - 1160.71.1170 Boehringer Ingelheim Investigational Site, Sassari
- Malaysia (2):
  - 1160.71.1291 Boehringer Ingelheim Investigational Site, Kuala Lumpur
  - 1160.71.1292 Boehringer Ingelheim Investigational Site, Kuala Lumpur
- Netherlands (27):
  - 1160.71.1337 Boehringer Ingelheim Investigational Site, 's-Hertogenbosch
  - 1160.71.1344 Boehringer Ingelheim Investigational Site, Almelo
  - 1160.71.1331 Boehringer Ingelheim Investigational Site, Amsterdam
  - 1160.71.1336 Boehringer Ingelheim Investigational Site, Apeldoorn
  - 1160.71.1332 Boehringer Ingelheim Investigational Site, Breda
  - 1160.71.1349 Boehringer Ingelheim Investigational Site, Den Helder
  - 1160.71.1345 Boehringer Ingelheim Investigational Site, Deventer
  - 1160.71.1360 Boehringer Ingelheim Investigational Site, Dirksland
  - 1160.71.1340 Boehringer Ingelheim Investigational Site, Ede
  - 1160.71.1358 Boehringer Ingelheim Investigational Site, Eindhoven
  - 1160.71.1338 Boehringer Ingelheim Investigational Site, Enschede
  - 1160.71.1343 Boehringer Ingelheim Investigational Site, Goes
  - 1160.71.1347 Boehringer Ingelheim Investigational Site, Gorinchem
  - 1160.71.1333 Boehringer Ingelheim Investigational Site, Groningen
  - 1160.71.1361 Boehringer Ingelheim Investigational Site, Heerlen
  - 1160.71.1339 Boehringer Ingelheim Investigational Site, Hengelo
  - 1160.71.1346 Boehringer Ingelheim Investigational Site, Hilversum
  - 1160.71.1356 Boehringer Ingelheim Investigational Site, Hoorn
  - 1160.71.1359 Boehringer Ingelheim Investigational Site, Maastricht
  - 1160.71.1341 Boehringer Ingelheim Investigational Site, Meppel
  - 1160.71.1354 Boehringer Ingelheim Investigational Site, Rotterdam
  - 1160.71.1351 Boehringer Ingelheim Investigational Site, Sneek
  - 1160.71.1353 Boehringer Ingelheim Investigational Site, Tiel
  - 1160.71.1352 Boehringer Ingelheim Investigational Site, Tilburg
  - 1160.71.1350 Boehringer Ingelheim Investigational Site, Veldhoven
  - 1160.71.1342 Boehringer Ingelheim Investigational Site, Velp
  - 1160.71.1348 Boehringer Ingelheim Investigational Site, Zwijndrecht
- Norway (6):
  - 1160.71.1396 Boehringer Ingelheim Investigational Site, Gjøvik
  - 1160.71.1393 Boehringer Ingelheim Investigational Site, Moss
  - 1160.71.1395 Boehringer Ingelheim Investigational Site, Nordbyhagen
  - 1160.71.1391 Boehringer Ingelheim Investigational Site, Oslo
  - 1160.71.1397 Boehringer Ingelheim Investigational Site, Oslo
  - 1160.71.1394 Boehringer Ingelheim Investigational Site, Rud
- Philippines (5):
  - 1160.71.1422 Boehringer Ingelheim Investigational Site, Ermita Manila
  - 1160.71.1421 Boehringer Ingelheim Investigational Site, Manila
  - 1160.71.1424 Boehringer Ingelheim Investigational Site, Pasig
  - 1160.71.1423 Boehringer Ingelheim Investigational Site, Quezon City
  - 1160.71.1425 Boehringer Ingelheim Investigational Site, Quezon City
- Poland (7):
  - 1160.71.1436 Boehringer Ingelheim Investigational Site, Gdynia
  - 1160.71.1437 Boehringer Ingelheim Investigational Site, Gdynia
  - 1160.71.1438 Boehringer Ingelheim Investigational Site, Gdynia
  - 1160.71.1433 Boehringer Ingelheim Investigational Site, Puławy
  - 1160.71.1431 Boehringer Ingelheim Investigational Site, Warsaw
  - 1160.71.1432 Boehringer Ingelheim Investigational Site, Warsaw
  - 1160.71.1434 Boehringer Ingelheim Investigational Site, Zabrze
- Portugal (6):
  - 1160.71.1456 Boehringer Ingelheim Investigational Site, Amadora
  - 1160.71.1451 Boehringer Ingelheim Investigational Site, Carnaxide
  - 1160.71.1454 Boehringer Ingelheim Investigational Site, Coimbra
  - 1160.71.1459 Boehringer Ingelheim Investigational Site, Coimbra
  - 1160.71.1457 Boehringer Ingelheim Investigational Site, Covilha
  - 1160.71.1455 Boehringer Ingelheim Investigational Site, Porto
- Romania (2):
  - 1160.71.1471 Boehringer Ingelheim Investigational Site, Bucharest
  - 1160.71.1472 Boehringer Ingelheim Investigational Site, Bucharest
- Russia (12):
  - 1160.71.1501 Boehringer Ingelheim Investigational Site, Moscow
  - 1160.71.1503 Boehringer Ingelheim Investigational Site, Moscow
  - 1160.71.1504 Boehringer Ingelheim Investigational Site, Moscow
  - 1160.71.1505 Boehringer Ingelheim Investigational Site, Moscow
  - 1160.71.1507 Boehringer Ingelheim Investigational Site, Moscow
  - 1160.71.1508 Boehringer Ingelheim Investigational Site, Moscow
  - 1160.71.1509 Boehringer Ingelheim Investigational Site, Moscow
  - 1160.71.1510 Boehringer Ingelheim Investigational Site, Moscow
  - 1160.71.1511 Boehringer Ingelheim Investigational Site, Moscow
  - 1160.71.1512 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1160.71.1513 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1160.71.1514 Boehringer Ingelheim Investigational Site, Saint Petersburg
- 1160.71.1531 Boehringer Ingelheim Investigational Site, Singapore, Singapore
- Slovakia (6):
  - 1160.71.1548 Boehringer Ingelheim Investigational Site, Banská Bystrica
  - 1160.71.1541 Boehringer Ingelheim Investigational Site, Bratislava
  - 1160.71.1542 Boehringer Ingelheim Investigational Site, Bratislava
  - 1160.71.1543 Boehringer Ingelheim Investigational Site, Bratislava
  - 1160.71.1550 Boehringer Ingelheim Investigational Site, Košice
  - 1160.71.1547 Boehringer Ingelheim Investigational Site, Žilina
- South Korea (11):
  - 1160.71.1585 Boehringer Ingelheim Investigational Site, Busan
  - 1160.71.1586 Boehringer Ingelheim Investigational Site, Cheonan-si
  - 1160.71.1584 Boehringer Ingelheim Investigational Site, Daegu
  - 1160.71.1591 Boehringer Ingelheim Investigational Site, Daegu
  - 1160.71.1590 Boehringer Ingelheim Investigational Site, Gwangju
  - 1160.71.1581 Boehringer Ingelheim Investigational Site, Incheon
  - 1160.71.1582 Boehringer Ingelheim Investigational Site, Seoul
  - 1160.71.1583 Boehringer Ingelheim Investigational Site, Seoul
  - 1160.71.1589 Boehringer Ingelheim Investigational Site, Seoul
  - 1160.71.1592 Boehringer Ingelheim Investigational Site, Seoul
  - 1160.71.1593 Boehringer Ingelheim Investigational Site, Seoul
- Sweden (11):
  - 1160.71.1633 Boehringer Ingelheim Investigational Site, Gothenburg
  - 1160.71.1627 Boehringer Ingelheim Investigational Site, Malmo
  - 1160.71.1628 Boehringer Ingelheim Investigational Site, Nässjö
  - 1160.71.1625 Boehringer Ingelheim Investigational Site, Norrköping
  - 1160.71.1623 Boehringer Ingelheim Investigational Site, Örebro
  - 1160.71.1626 Boehringer Ingelheim Investigational Site, Stockholm
  - 1160.71.1634 Boehringer Ingelheim Investigational Site, Stockholm
  - 1160.71.1624 Boehringer Ingelheim Investigational Site, Umeå
  - 1160.71.1621 Boehringer Ingelheim Investigational Site, Uppsala
  - 1160.71.1635 Boehringer Ingelheim Investigational Site, Uppsala
  - 1160.71.1622 Boehringer Ingelheim Investigational Site, Västerås
- Switzerland (4):
  - 1160.71.1652 Boehringer Ingelheim Investigational Site, Basel
  - 1160.71.1655 Boehringer Ingelheim Investigational Site, Bellinzona
  - 1160.71.1651 Boehringer Ingelheim Investigational Site, Bern
  - 1160.71.1654 Boehringer Ingelheim Investigational Site, Lugano
- Taiwan (13):
  - 1160.71.1680 Boehringer Ingelheim Investigational Site, Changhua
  - 1160.71.1683 Boehringer Ingelheim Investigational Site, Hualien City
  - 1160.71.1682 Boehringer Ingelheim Investigational Site, Kaohsiung City
  - 1160.71.1679 Boehringer Ingelheim Investigational Site, Taichung
  - 1160.71.1681 Boehringer Ingelheim Investigational Site, Tainan
  - 1160.71.1671 Boehringer Ingelheim Investigational Site, Taipei
  - 1160.71.1672 Boehringer Ingelheim Investigational Site, Taipei
  - 1160.71.1673 Boehringer Ingelheim Investigational Site, Taipei
  - 1160.71.1674 Boehringer Ingelheim Investigational Site, Taipei
  - 1160.71.1675 Boehringer Ingelheim Investigational Site, Taipei
  - 1160.71.1676 Boehringer Ingelheim Investigational Site, Taipei
  - 1160.71.1677 Boehringer Ingelheim Investigational Site, Taipei
  - 1160.71.1678 Boehringer Ingelheim Investigational Site, Taoyuan District
- Thailand (3):
  - 1160.71.1701 Boehringer Ingelheim Investigational Site, Bangkok
  - 1160.71.1703 Boehringer Ingelheim Investigational Site, Chiang Mai
  - 1160.71.1704 Boehringer Ingelheim Investigational Site, Khon Kaen
- United Kingdom (10):
  - 1160.71.1744 Boehringer Ingelheim Investigational Site, Birmingham
  - 1160.71.1746 Boehringer Ingelheim Investigational Site, Chertsey
  - 1160.71.1745 Boehringer Ingelheim Investigational Site, County Armagh
  - 1160.71.1755 Boehringer Ingelheim Investigational Site, Kirkcaldy, Fife
  - 1160.71.1741 Boehringer Ingelheim Investigational Site, London
  - 1160.71.1742 Boehringer Ingelheim Investigational Site, Newcastle upon Tyne
  - 1160.71.1751 Boehringer Ingelheim Investigational Site, Newport
  - 1160.71.1752 Boehringer Ingelheim Investigational Site, Northampton
  - 1160.71.1743 Boehringer Ingelheim Investigational Site, Romford, Essex
  - 1160.71.1748 Boehringer Ingelheim Investigational Site, York

REFERENCES:
- [Derived] Connolly SJ, Wallentin L, Ezekowitz MD, Eikelboom J, Oldgren J, Reilly PA, Brueckmann M, Pogue J, Alings M, Amerena JV, Avezum A, Baumgartner I, Budaj AJ, Chen JH, Dans AL, Darius H, Di Pasquale G, Ferreira J, Flaker GC, Flather MD, Franzosi MG, Golitsyn SP, Halon DA, Heidbuchel H, Hohnloser SH, Huber K, Jansky P, Kamensky G, Keltai M, Kim SS, Lau CP, Le Heuzey JY, Lewis BS, Liu L, Nanas J, Omar R, Pais P, Pedersen KE, Piegas LS, Raev D, Smith PJ, Talajic M, Tan RS, Tanomsup S, Toivonen L, Vinereanu D, Xavier D, Zhu J, Wang SQ, Duffy CO, Themeles E, Yusuf S. The Long-Term Multicenter Observational Study of Dabigatran Treatment in Patients With Atrial Fibrillation (RELY-ABLE) Study. Circulation. 2013 Jul 16;128(3):237-43. doi: 10.1161/CIRCULATIONAHA.112.001139. Epub 2013 Jun 14. PMID 23770747

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 5897 subjects were enrolled (rolled over from RE-LY trial), and 5891 were entered in this study. There were 8 subjects not treated; therefore 5883 subjects comprise the 'started' treatment group.
Groups:
- Dabigatran 110 mg: Dabigatran etexilate 110 mg twice daily
- Dabigatran 150 mg: Dabigatran etexilate 150 mg twice daily
Period: Overall Study
Arm/Group | Dabigatran 110 mg | Dabigatran 150 mg
Started | 2927 (Number of patients which are treated.) | 2956 (Number of patients which are treated.)
Completed | 2446 | 2438
Not Completed | 481 | 518
Not completed — Major/minor bleed | 30 | 44
Not completed — Outcome event - other | 33 | 25
Not completed — Adverse Event | 111 | 121
Not completed — Hospitalization (not including surgery) | 18 | 17
Not completed — Hospitalization due to surgery | 37 | 40
Not completed — Reduced creatinine clearance | 53 | 55
Not completed — Elevated LFT results | 7 | 3
Not completed — Patient refused to take study medication | 65 | 76
Not completed — Missing | 1 | 0
Not completed — Death | 1 | 1
Not completed — Procedure | 6 | 7
Not completed — Withdrawal by Subject | 21 | 25
Not completed — Site closed | 4 | 3
Not completed — Physician Decision | 47 | 38
Not completed — Protocol Violation | 3 | 11
Not completed — Patient elected | 7 | 9
Not completed — Site closed for cause | 19 | 19
Not completed — Other reason not defined above | 5 | 5
Not completed — Excluded from analysis | 13 | 19

BASELINE CHARACTERISTICS:
Population: SAF - Safety set; included all treated subjects, but excluded subjects from sites 1059 and 0246.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dabigatran 110 mg | Dabigatran 150 mg | Total
Number analyzed (Participants) | 2914 | 2937 | 5851
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.1 (8.4) | 73.1 (8.4) | 73.1 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1000 | 1026 | 2026
  Male | 1914 | 1911 | 3825

OUTCOME MEASURES:

1. Primary Outcome: Major Bleeding, Annualized Rate of Subjects With Major Bleeds
Description: Annualized event rate (%) = 100 * No. subjects with event / subject-years. Subject-years = Sum (date of last visit - date of first dose + 1) of all subjects / 365.25.
  Major bleeding must have satisfied one or more of the following criteria:
  * Bleeding associated with a reduction in hemoglobin of at least 20 g/L
  * Required transfusion of at least 2 units of blood or packed cells
  * Symptomatic bleeding in a critical area or organ: intraocular, intraspinal, intramuscular with compartment syndrome, retroperitoneal, intra-articular, pericardial, gastrointestinal
  Major bleed were classified as life-threatening if they met one or more of the following criteria:
  * Reduction in hemoglobin of at least 50 g/L
  * Transfusion of at least 4 units of blood or packed cells
  * Symptomatic intracranial bleeding, either subdural or intracerebral
  * Associated with hypotension requiring use of intravenous inotropic agents
  * Required surgical intervention to stop bleeding
  * Resulted in death
Time Frame: up to 43 months
Population: SAF-FAS interval
Measure: Number; unit: percentage of subject-years
Arm/Group | Dabigatran 110 mg | Dabigatran 150 mg
Number analyzed (Participants) | 2914 | 2937
percentage of subject-years | 2.79 | 3.59
Statistical Analysis 1: Comparison: Dabigatran 110 mg vs Dabigatran 150 mg; Test type: Superiority or Other; p = 0.0055, Regression, Cox; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.64 to 0.93]

2. Secondary Outcome: Stroke, Annualized Rate of Subjects With Stroke
Description: Annualized event rate (%) = 100 * No. subjects with event / subject-years. Subject-years = Sum (date of last visit - date of first dose + 1) of all subjects / 365.25.
  Stroke was an acute onset of a focal neurological deficit of presumed vascular origin lasting for 24 hours or more or resulting in death. The stroke was categorized as ischemic or hemorrhagic or cause unknown based on computerized tomography (CT), magnetic resonance (MR) scanning or autopsy. Fatal stroke was defined as death from any cause within 30 days of stroke. Severity of stroke was assessed by modified Rankin score at discharge from hospital
Time Frame: up to 43 months
Population: SAF-FAS interval
Measure: Number; unit: percentage of subject-years
Arm/Group | Dabigatran 110 mg | Dabigatran 150 mg
Number analyzed (Participants) | 2914 | 2937
percentage of subject-years | 1.39 | 1.26

3. Secondary Outcome: Non CNS Systemic Embolism (SEE), Annualized Rate of Subjects With Non-CNS SEE
Description: Annualized event rate (%) = 100 * No. subjects with event / subject-years. Subject-years = Sum (date of last visit - date of first dose + 1) of all subjects / 365.25.
  Systemic embolism was an acute vascular occlusion of the extremities or any organ (kidneys, mesenteric arteries, spleen, retina or grafts), and was to be documented by angiography, surgery, scintigraphy, or autopsy.
Time Frame: up to 43 months
Population: SAF-FAS interval
Measure: Number; unit: percentage of subject-years
Arm/Group | Dabigatran 110 mg | Dabigatran 150 mg
Number analyzed (Participants) | 2914 | 2937
percentage of subject-years | 0.25 | 0.23

4. Secondary Outcome: Pulmonary Embolism (PE), Annualized Rate of Subjects With PE
Description: Annualized event rate (%) = 100 * No. subjects with event / subject-years. Subject-years = Sum (date of last visit - date of first dose + 1) of all subjects / 365.25.
  Pulmonary Embolism was generally documented by one of the following:
  1. an intraluminal filling defect in segmental or more proximal branches on spiral CT scan
  2. an intraluminal filling defect or an extension of an existing defect or a sudden cutoff of vessels more than 2.5 mm in diameter on the pulmonary angiogram
  3. a perfusion defect of at least 75% of a segment with a local normal ventilation result (high-probability) on ventilation/perfusion lung scan (VPLS)
  4. inconclusive spiral CT, pulmonary angiography or lung scintigraphy with demonstration of DVT in the lower extremities by compression ultrasound or venography.
Time Frame: up to 43 months
Population: SAF-FAS interval
Measure: Number; unit: percentage of subject-years
Arm/Group | Dabigatran 110 mg | Dabigatran 150 mg
Number analyzed (Participants) | 2914 | 2937
percentage of subject-years | 0.10 | 0.12

5. Secondary Outcome: Acute Myocardial Infarction (MI), Annualized Rate of Subjects With MI
Description: Annualized event rate (%) = 100 * No. subjects with event / subject-years. Subject-years = Sum (date of last visit - date of first dose + 1) of all subjects / 365.25.
  a. In subjects not undergoing PCI or CABG a subject should have fulfilled at least 2 of the following: i. Typical prolonged severe chest pain or related symptoms or signs suggestive of MI. ii. Elevation of troponin or CK-MB to more than upper level of normal (ULN) or, if CK-MB was elevated at baseline, re-elevation to more than 50% increase above the previous level. iii. Development of significant Q-waves in at least 2 adjacent ECG leads. b. After percutaneous coronary intervention (within 24h). c. After coronary artery bypass grafting (within 72h). d. Silent myocardial infarction. e. Myocardial infarction could also have been demonstrated at autopsy.
Time Frame: up to 43 months
Population: SAF-FAS interval
Measure: Number; unit: percentage of subject-years
Arm/Group | Dabigatran 110 mg | Dabigatran 150 mg
Number analyzed (Participants) | 2914 | 2937
percentage of subject-years | 0.72 | 0.66

6. Secondary Outcome: Deep Vein Thrombosis, Annualized Rate of Subjects With DVT
Description: Annualized event rate (%) = 100 * No. subjects with event / subject-years. Subject-years = Sum (date of last visit - date of first dose + 1) of all subjects / 365.25.
  Deep Vein Thrombosis (DVT) was generally documented by one of the following:
  1. abnormal compression ultrasound (CUS),
  2. an intraluminal filling defect on venography.
Time Frame: up to 43 months
Population: SAF-FAS interval
Measure: Number; unit: percentage of subject-years
Arm/Group | Dabigatran 110 mg | Dabigatran 150 mg
Number analyzed (Participants) | 2914 | 2937
percentage of subject-years | 0.06 | 0.11

7. Secondary Outcome: Death, Annualized Rate of Subject Death
Description: Annualized event rate (%) = 100 * No. subjects with event / subject-years. Subject-years = Sum (date of last visit - date of first dose + 1) of all subjects / 365.25.
  Deaths were classified as being vascular (sudden/arrhythmic, pump failure death, or other vascular, including bleeding) or non-vascular, due to other specified causes (e.g., malignancy), or of unknown etiology.
Time Frame: up to 43 months
Population: SAF-FAS interval
Measure: Number; unit: percentage of subject-years
Arm/Group | Dabigatran 110 mg | Dabigatran 150 mg
Number analyzed (Participants) | 2914 | 2937
percentage of subject-years | 3.18 | 2.99

8. Secondary Outcome: Annualized Rate of Subjects With Composite Incidence of Stroke, Non CNS Systemic Embolism (SEE)
Description: Annualized event rate (%) = 100 * No. subjects with event / subject-years. Subject-years = Sum (date of last visit - date of first dose + 1) of all subjects / 365.25.
Time Frame: up to 43 months
Population: SAF-FAS interval
Measure: Number; unit: percentage of subject-years
Arm/Group | Dabigatran 110 mg | Dabigatran 150 mg
Number analyzed (Participants) | 2914 | 2937
percentage of subject-years | 1.60 | 1.47
Statistical Analysis 1: Comparison: Dabigatran 110 mg vs Dabigatran 150 mg; Test type: Superiority or Other; p = 0.5119, Regression, Cox; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.84 to 1.42]

9. Secondary Outcome: Annualized Rate of Subjects With Composite Incidence of Stroke, Non CNS Systemic Embolism (SEE) and All Cause Death
Description: as for outcome 8
Time Frame: up to 43 months
Population: SAF-FAS interval
Measure: Number; unit: percentage of subject-years
Arm/Group | Dabigatran 110 mg | Dabigatran 150 mg
Number analyzed (Participants) | 2914 | 2937
percentage of subject-years | 4.40 | 4.02
Statistical Analysis 1: Comparison: Dabigatran 110 mg vs Dabigatran 150 mg; Test type: Superiority or Other; p = 0.2371, Regression, Cox; Hazard Ratio (HR) = 1.10, 95% CI 2-sided [0.94 to 1.29]

10. Secondary Outcome: Annualized Rate of Subjects With Composite Incidence of Stroke, Non CNS Systemic Embolism (SEE), Pulmonary Embolism (PE), Myocardial Infarction, Vascular Death
Description: as for outcome 8
Time Frame: up to 43 months
Population: SAF-FAS interval
Measure: Number; unit: percentage of subject-years
Arm/Group | Dabigatran 110 mg | Dabigatran 150 mg
Number analyzed (Participants) | 2914 | 2937
percentage of subject-years | 3.51 | 3.32
Statistical Analysis 1: Comparison: Dabigatran 110 mg vs Dabigatran 150 mg; Test type: Superiority or Other; p = 0.5052, Regression, Cox; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.89 to 1.27]

11. Secondary Outcome: Annualized Rate of Subjects With Composite Incidence of Stroke, Non CNS Systemic Embolism (SEE), Pulmonary Embolism (PE), Myocardial Infarction (MI), All Cause Death and Major Bleed
Description: as for outcome 8
Time Frame: up to 43 months
Population: SAF-FAS interval
Measure: Number; unit: percentage of subject-years
Arm/Group | Dabigatran 110 mg | Dabigatran 150 mg
Number analyzed (Participants) | 2914 | 2937
percentage of subject-years | 6.65 | 7.14
Statistical Analysis 1: Comparison: Dabigatran 110 mg vs Dabigatran 150 mg; Test type: Superiority or Other; p = 0.2241, Regression, Cox; Hazard Ratio (HR) = 0.93, 95% CI [0.82 to 1.05]

12. Secondary Outcome: Annualized Rate of Subjects With Minor Bleeds
Description: Annualized event rate (%) = 100 * No. subjects with event / subject-years. Subject-years = Sum (date of last visit - date of first dose + 1) of all subjects / 365.25.
  Minor bleeds were clinical bleeds that did not fulfill the criteria for major bleeds. Minor bleeds were classified as associated with study medication discontinuation (temporary or permanent) or not.
Time Frame: up to 43 months
Population: SAF-FAS interval
Measure: Number; unit: percentage of subject-years
Arm/Group | Dabigatran 110 mg | Dabigatran 150 mg
Number analyzed (Participants) | 2914 | 2937
percentage of subject-years | 7.49 | 8.98

13. Secondary Outcome: Annualized Rate of Subjects With Any Bleeds (Major Plus Minor)
Description: as for outcome 8
Time Frame: up to 43 months
Population: SAF-FAS interval
Measure: Number; unit: percentage of subject-years
Arm/Group | Dabigatran 110 mg | Dabigatran 150 mg
Number analyzed (Participants) | 2914 | 2937
percentage of subject-years | 9.44 | 11.20

14. Secondary Outcome: Annualized Rate of Subjects With Intra-Cranial Hemorrhage (ICH)
Description: as for outcome 8
Time Frame: up to 43 months
Population: SAF-FAS interval
Measure: Number; unit: percentage of subject-years
Arm/Group | Dabigatran 110 mg | Dabigatran 150 mg
Number analyzed (Participants) | 2914 | 2937
percentage of subject-years | 0.28 | 0.33

ADVERSE EVENTS:
Time Frame: Up to 43 months
Arm/Group | Dabigatran 110 mg | Dabigatran 150 mg
Serious Adverse Events (participants affected / at risk) | 1028/2914 | 1106/2937
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran 110 mg (N=2914) | Dabigatran 150 mg (N=2937)
Anaemia (Blood and lymphatic system disorders) | 23 | 36
Coagulopathy (Blood and lymphatic system disorders) | 1 | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 4
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 4 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Polycythaemia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 5
Acute coronary syndrome (Cardiac disorders) | 2 | 6
Acute left ventricular failure (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 34 | 36
Angina unstable (Cardiac disorders) | 2 | 13
Aortic valve stenosis (Cardiac disorders) | 1 | 1
Arrhythmia (Cardiac disorders) | 5 | 4
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 2
Atrial fibrillation (Cardiac disorders) | 84 | 95
Atrial flutter (Cardiac disorders) | 4 | 6
Atrial tachycardia (Cardiac disorders) | 1 | 1
Atrial thrombosis (Cardiac disorders) | 1 | 2
Atrioventricular block (Cardiac disorders) | 1 | 1
Atrioventricular block complete (Cardiac disorders) | 2 | 4
Bradyarrhythmia (Cardiac disorders) | 3 | 6
Bradycardia (Cardiac disorders) | 19 | 23
Cardiac arrest (Cardiac disorders) | 7 | 9
Cardiac failure (Cardiac disorders) | 70 | 87
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 3 | 3
Cardiac failure congestive (Cardiac disorders) | 68 | 71
Cardiac valve disease (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 2 | 2
Cardiogenic shock (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 2
Chronotropic incompetence (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 14 | 12
Coronary artery occlusion (Cardiac disorders) | 0 | 2
Coronary artery stenosis (Cardiac disorders) | 0 | 2
Dressler's syndrome (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 3
Left ventricular failure (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 7 | 5
Mitral valve stenosis (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 3 | 2
Myocardial ischaemia (Cardiac disorders) | 3 | 1
Palpitations (Cardiac disorders) | 4 | 5
Pericardial effusion (Cardiac disorders) | 3 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Right ventricular failure (Cardiac disorders) | 1 | 2
Sick sinus syndrome (Cardiac disorders) | 13 | 10
Sinus arrest (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 2 | 5
Tricuspid valve incompetence (Cardiac disorders) | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 7 | 8
Ventricular fibrillation (Cardiac disorders) | 4 | 6
Ventricular tachycardia (Cardiac disorders) | 7 | 6
Deafness (Ear and labyrinth disorders) | 0 | 2
Hearing impaired (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 6 | 4
Vertigo positional (Ear and labyrinth disorders) | 2 | 0
Addison's disease (Endocrine disorders) | 0 | 1
Goitre (Endocrine disorders) | 1 | 1
Hyperparathyroidism (Endocrine disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 2 | 0
Amaurosis fugax (Eye disorders) | 1 | 0
Blepharochalasis (Eye disorders) | 0 | 1
Blindness (Eye disorders) | 1 | 0
Cataract (Eye disorders) | 8 | 10
Diplopia (Eye disorders) | 1 | 0
Eye haemorrhage (Eye disorders) | 0 | 2
Glaucoma (Eye disorders) | 1 | 0
Macular pseudohole (Eye disorders) | 0 | 1
Optic ischaemic neuropathy (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 2 | 0
Retinal haemorrhage (Eye disorders) | 0 | 1
Retinal vein occlusion (Eye disorders) | 1 | 1
Scotoma (Eye disorders) | 1 | 0
Ulcerative keratitis (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 1
Abdominal mass (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 29 | 27
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 2
Colitis ischaemic (Gastrointestinal disorders) | 1 | 1
Colonic obstruction (Gastrointestinal disorders) | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 11 | 4
Constipation (Gastrointestinal disorders) | 2 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 8 | 3
Diverticulum (Gastrointestinal disorders) | 0 | 3
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 2
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 3
Duodenal polyp (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 4 | 4
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 7 | 12
Dysphagia (Gastrointestinal disorders) | 3 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 2
Gastric ulcer (Gastrointestinal disorders) | 8 | 5
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 8 | 7
Gastritis erosive (Gastrointestinal disorders) | 0 | 2
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 4
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 20 | 20
Gastrointestinal mucosal disorder (Gastrointestinal disorders) | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 3 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 2
Hiatus hernia (Gastrointestinal disorders) | 0 | 2
Ileus (Gastrointestinal disorders) | 6 | 7
Inguinal hernia (Gastrointestinal disorders) | 13 | 7
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 2 | 3
Intestinal obstruction (Gastrointestinal disorders) | 8 | 2
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Large intestinal ulcer (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 6
Melaena (Gastrointestinal disorders) | 6 | 5
Mesenteric artery stenosis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 1
Obstruction gastric (Gastrointestinal disorders) | 1 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 2
Oesophageal achalasia (Gastrointestinal disorders) | 0 | 1
Oesophageal obstruction (Gastrointestinal disorders) | 0 | 1
Oesophageal rupture (Gastrointestinal disorders) | 0 | 1
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 3
Oesophagitis (Gastrointestinal disorders) | 0 | 2
Pancreatic cyst (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 4
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 5 | 5
Rectal prolapse (Gastrointestinal disorders) | 1 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 5 | 6
Subileus (Gastrointestinal disorders) | 1 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 5
Vomiting (Gastrointestinal disorders) | 6 | 6
Adverse drug reaction (General disorders) | 1 | 1
Asthenia (General disorders) | 7 | 10
Chest discomfort (General disorders) | 2 | 1
Chest pain (General disorders) | 35 | 47
Death (General disorders) | 1 | 1
Device breakage (General disorders) | 1 | 0
Device dislocation (General disorders) | 3 | 1
Device malfunction (General disorders) | 1 | 1
Drug ineffective (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Gait disturbance (General disorders) | 2 | 0
General physical health deterioration (General disorders) | 1 | 3
Generalised oedema (General disorders) | 0 | 1
Hernia (General disorders) | 6 | 4
Hernia obstructive (General disorders) | 1 | 0
Impaired healing (General disorders) | 2 | 1
Malaise (General disorders) | 1 | 1
Medical device complication (General disorders) | 0 | 1
Multi-organ disorder (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 3 | 2
Necrosis (General disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 5 | 3
Oedema (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 5 | 4
Pain (General disorders) | 1 | 1
Pyrexia (General disorders) | 3 | 4
Stent-graft endoleak (General disorders) | 0 | 1
Sudden cardiac death (General disorders) | 1 | 0
Sudden death (General disorders) | 0 | 2
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 4 | 1
Biliary colic (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 4 | 1
Cholangitis acute (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 10 | 7
Cholecystitis acute (Hepatobiliary disorders) | 4 | 0
Cholelithiasis (Hepatobiliary disorders) | 10 | 4
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 1
Hepatitis toxic (Hepatobiliary disorders) | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 1
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 1
Anaphylactic shock (Immune system disorders) | 1 | 0
Abscess (Infections and infestations) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 2
Abscess neck (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 3 | 3
Arthritis bacterial (Infections and infestations) | 2 | 1
Arthritis infective (Infections and infestations) | 0 | 2
Atypical pneumonia (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 4 | 1
Brain abscess (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 11 | 8
Bronchitis viral (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 2 | 1
Cellulitis (Infections and infestations) | 25 | 25
Cellulitis staphylococcal (Infections and infestations) | 1 | 0
Cholecystitis infective (Infections and infestations) | 2 | 1
Chronic sinusitis (Infections and infestations) | 1 | 0
Clostridial infection (Infections and infestations) | 3 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 2
Corneal abscess (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 2 | 1
Dengue fever (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 3
Diabetic foot infection (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 6
Ear infection (Infections and infestations) | 1 | 1
Endocarditis (Infections and infestations) | 5 | 1
Endocarditis bacterial (Infections and infestations) | 0 | 1
Enterococcal sepsis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 7 | 6
Escherichia sepsis (Infections and infestations) | 1 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 2
Eye infection (Infections and infestations) | 0 | 1
Fungal infection (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 2 | 2
Gastric ulcer helicobacter (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 3 | 4
Gastroenteritis cryptosporidial (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 2
Gastrointestinal infection (Infections and infestations) | 1 | 0
Groin abscess (Infections and infestations) | 1 | 0
Groin infection (Infections and infestations) | 0 | 1
Herpes ophthalmic (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 4
Herpes zoster ophthalmic (Infections and infestations) | 0 | 1
Herpes zoster oticus (Infections and infestations) | 0 | 1
Implant site infection (Infections and infestations) | 2 | 1
Infected bites (Infections and infestations) | 0 | 1
Infected cyst (Infections and infestations) | 1 | 0
Infected skin ulcer (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 5 | 5
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 1 | 2
Klebsiella sepsis (Infections and infestations) | 1 | 0
Labyrinthitis (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 2 | 0
Lobar pneumonia (Infections and infestations) | 3 | 3
Localised infection (Infections and infestations) | 4 | 5
Lower respiratory tract infection (Infections and infestations) | 2 | 2
Lung infection (Infections and infestations) | 0 | 2
Nasopharyngitis (Infections and infestations) | 0 | 1
Neuroborreliosis (Infections and infestations) | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 1 | 0
Oesophageal infection (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 2
Osteomyelitis (Infections and infestations) | 2 | 4
Otitis externa (Infections and infestations) | 0 | 1
Pancreatic abscess (Infections and infestations) | 0 | 1
Parotitis (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 1 | 1
Peritonitis bacterial (Infections and infestations) | 1 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 1
Pharyngeal abscess (Infections and infestations) | 1 | 0
Pharyngolaryngeal abscess (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 91 | 99
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pneumonia legionella (Infections and infestations) | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 3 | 2
Postoperative wound infection (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 3
Pyelonephritis acute (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 5 | 3
Sepsis (Infections and infestations) | 19 | 23
Septic shock (Infections and infestations) | 2 | 1
Sinusitis (Infections and infestations) | 1 | 1
Skin infection (Infections and infestations) | 2 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Staphylococcal skin infection (Infections and infestations) | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 5 | 5
Urethritis chlamydial (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 21 | 29
Urinary tract infection bacterial (Infections and infestations) | 0 | 1
Urinary tract infection pseudomonal (Infections and infestations) | 1 | 0
Urinary tract infection staphylococcal (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 3 | 2
Viral infection (Infections and infestations) | 1 | 3
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 3 | 8
Arterial injury (Injury, poisoning and procedural complications) | 1 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 | 0
Cartilage injury (Injury, poisoning and procedural complications) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 3 | 2
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Deafness traumatic (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 26 | 31
Fat embolism (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 4 | 9
Femur fracture (Injury, poisoning and procedural complications) | 10 | 6
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 3 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 2
Hip fracture (Injury, poisoning and procedural complications) | 11 | 11
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 1
Iatrogenic injury (Injury, poisoning and procedural complications) | 1 | 0
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 2
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 2
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 2
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 3 | 3
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0
Open wound (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 4 | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Procedural hypertension (Injury, poisoning and procedural complications) | 0 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 3
Radius fracture (Injury, poisoning and procedural complications) | 1 | 3
Rib fracture (Injury, poisoning and procedural complications) | 3 | 3
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 4
Skin injury (Injury, poisoning and procedural complications) | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0
Snake bite (Injury, poisoning and procedural complications) | 1 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 2 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 5 | 5
Sternal fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 5 | 4
Subdural haemorrhage (Injury, poisoning and procedural complications) | 2 | 2
Tendon injury (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 2 | 3
Toxicity to various agents (Injury, poisoning and procedural complications) | 5 | 1
Traumatic arthritis (Injury, poisoning and procedural complications) | 0 | 1
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 3
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 3
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Wound necrosis (Injury, poisoning and procedural complications) | 3 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 2 | 2
Blood glucagon abnormal (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 0 | 1
Creatinine renal clearance decreased (Investigations) | 2 | 2
Haemoglobin decreased (Investigations) | 5 | 0
Heart rate decreased (Investigations) | 2 | 0
Heart rate irregular (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 3 | 1
International normalised ratio increased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 2 | 2
Platelet count decreased (Investigations) | 0 | 1
Troponin I increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 2 | 2
Dehydration (Metabolism and nutrition disorders) | 11 | 20
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 3 | 2
Diabetic complication (Metabolism and nutrition disorders) | 0 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 2
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 4 | 6
Haemochromatosis (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 8 | 8
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 2
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 7
Arthritis (Musculoskeletal and connective tissue disorders) | 7 | 5
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 15
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 1
Crystal arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 2
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 4
Jaw cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 3
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 8
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 28 | 36
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 2
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 2 | 0
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 3
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 | 2
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 9
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bone neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bone sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 9
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Choroid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 | 6
Colon cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrooesophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Langerhans' cell histiocytosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Large cell carcinoma of the respiratory tract stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 16 | 5
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 5
Malignant neoplasm of pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Metastases to pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 5
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 | 14
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Rectal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Amnesia (Nervous system disorders) | 1 | 0
Aphasia (Nervous system disorders) | 1 | 0
Brachial plexopathy (Nervous system disorders) | 1 | 0
Brain stem stroke (Nervous system disorders) | 1 | 0
Carotid artery insufficiency (Nervous system disorders) | 1 | 0
Carotid artery occlusion (Nervous system disorders) | 1 | 1
Carotid artery stenosis (Nervous system disorders) | 4 | 5
Carotid sinus syndrome (Nervous system disorders) | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 1 | 1
Cerebellar haemorrhage (Nervous system disorders) | 2 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 2 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 8 | 5
Cervical root pain (Nervous system disorders) | 1 | 0
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 2 | 1
Coma (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 5 | 2
Dementia (Nervous system disorders) | 2 | 3
Dementia Alzheimer's type (Nervous system disorders) | 1 | 2
Dizziness (Nervous system disorders) | 4 | 7
Embolic stroke (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 4 | 2
Epilepsy (Nervous system disorders) | 2 | 1
Grand mal convulsion (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 2 | 1
Haemorrhagic stroke (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 3
Hemiparesis (Nervous system disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 2
IIIrd nerve paralysis (Nervous system disorders) | 1 | 0
Intraventricular haemorrhage (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 5 | 2
Lumbar radiculopathy (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Myasthenia gravis (Nervous system disorders) | 1 | 0
Myelopathy (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Normal pressure hydrocephalus (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 3 | 0
Paresis cranial nerve (Nervous system disorders) | 1 | 0
Parkinson's disease (Nervous system disorders) | 2 | 1
Parkinsonism (Nervous system disorders) | 2 | 1
Partial seizures (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 1 | 1
Presyncope (Nervous system disorders) | 1 | 4
Sciatic nerve palsy (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 1 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 2 | 1
Syncope (Nervous system disorders) | 24 | 24
Transient ischaemic attack (Nervous system disorders) | 6 | 4
Tremor (Nervous system disorders) | 0 | 1
Trigeminal neuralgia (Nervous system disorders) | 1 | 0
VIIth nerve paralysis (Nervous system disorders) | 2 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 2 | 0
Vertigo CNS origin (Nervous system disorders) | 0 | 1
Abnormal behaviour (Psychiatric disorders) | 1 | 0
Alcohol abuse (Psychiatric disorders) | 1 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 2 | 2
Delirium (Psychiatric disorders) | 3 | 2
Depression (Psychiatric disorders) | 1 | 5
Disorientation (Psychiatric disorders) | 0 | 1
Mental disorder (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 5 | 1
Panic attack (Psychiatric disorders) | 1 | 0
Panic disorder (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Bladder obstruction (Renal and urinary disorders) | 1 | 0
Bladder prolapse (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Glomerulonephritis (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 2 | 7
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 4 | 1
Nephrotic syndrome (Renal and urinary disorders) | 1 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 3
Renal cyst (Renal and urinary disorders) | 1 | 0
Renal disorder (Renal and urinary disorders) | 1 | 0
Renal embolism (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 19 | 9
Renal failure acute (Renal and urinary disorders) | 23 | 23
Renal failure chronic (Renal and urinary disorders) | 1 | 2
Renal impairment (Renal and urinary disorders) | 1 | 2
Renal infarct (Renal and urinary disorders) | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 3
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 12 | 13
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Pelvic haematoma (Reproductive system and breast disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Spermatocele (Reproductive system and breast disorders) | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Vaginal prolapse (Reproductive system and breast disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 27 | 30
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 34 | 32
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 11 | 7
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 2 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 | 0
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Activities of daily living impaired (Social circumstances) | 1 | 1
Dental implantation (Surgical and medical procedures) | 0 | 1
Lesion excision (Surgical and medical procedures) | 1 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 1
Aneurysm (Vascular disorders) | 0 | 1
Aortic aneurysm (Vascular disorders) | 11 | 8
Aortic aneurysm rupture (Vascular disorders) | 2 | 0
Aortic dissection (Vascular disorders) | 5 | 1
Aortic intramural haematoma (Vascular disorders) | 1 | 0
Aortic stenosis (Vascular disorders) | 6 | 6
Arteriosclerosis (Vascular disorders) | 0 | 3
Arteritis (Vascular disorders) | 0 | 1
Blood pressure inadequately controlled (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 2 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 6
Femoral artery aneurysm (Vascular disorders) | 1 | 0
Femoral artery occlusion (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 2 | 3
Haemorrhage (Vascular disorders) | 4 | 5
Hypertension (Vascular disorders) | 11 | 10
Hypertensive crisis (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 8 | 9
Intermittent claudication (Vascular disorders) | 1 | 2
Ischaemia (Vascular disorders) | 0 | 1
Leriche syndrome (Vascular disorders) | 1 | 1
Malignant hypertension (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 2 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 4 | 2
Peripheral artery aneurysm (Vascular disorders) | 1 | 0
Peripheral artery stenosis (Vascular disorders) | 2 | 4
Peripheral artery thrombosis (Vascular disorders) | 1 | 0
Peripheral embolism (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 2 | 1
Peripheral vascular disorder (Vascular disorders) | 2 | 4
Shock haemorrhagic (Vascular disorders) | 0 | 1
Temporal arteritis (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0
Venous occlusion (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Non-serious adverse events were not collected on subjects in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.